CLINICAL TRIAL: NCT01196338
Title: Early Weightbearing and Mobilization Versus Non-Weightbearing and Immobilization After ORIF of Unstable Ankle Fractures: a Randomized Controlled Trial
Brief Title: Early Weightbearing and Mobilization Versus Non-Weightbearing and Mobilization in Unstable Ankle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Orthopaedic Trauma Association (Other); Canadian Orthopaedic Foundation (Other); Künzli SwissSchuh (Unknown)
Responsible Party: Dr. Richard Jenkinson, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ankle
Record Dates: First submitted 2010-09-01; First posted 2010-09-08 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2010-09

CONDITIONS: Ankle Injuries
Keywords: Ankle fracture; Return to work; Return to function; Rehabilitation; Weight-bearing
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-weightbearing no ROM (Active Comparator): Patients will be placed in a back slab post-op and will remain non-weight bearing with crutches with no range of motion for a total of 6 weeks.
  After 6 weeks post-op, they will be placed in a boot orthosis and permitted to weight-bear as tolerated.
  Interventions: Behavioral: non-weight bearing, no range of motion
- Early weight-bearing and ROM (Experimental): Patients will be placed in a back slab post-operatively. At 2 weeks post op they will have the back slab removed and placed in a boot orthosis. At this time they will be permitted to weight-bear as tolerated and perform limited ankle range of motion exercises.
  After 6 weeks post op they will start to wean from the boot orthosis.
  Interventions: Behavioral: Early weight-bearing and range of motion exercises

INTERVENTIONS:
Behavioral: Early weight-bearing and range of motion exercises — * 0 weeks to 2 weeks: Posterior plaster slab or cast, non-weightbearing, crutches;
  * At 2 week visit to clinic: Posterior plaster slab or cast removed, staples/stitches removed placed in orthosis, with instructions to be weightbearing as tolerated. Instructions for limited range of motion to be given;
  * At 2 weeks to 6 weeks: Weightbearing as tolerated in orthosis, follow range of motion instructions;
  * After 6 weeks: Instructions to continue weightbearing as tolerated, wean from orthosis.
  Arms: Early weight-bearing and ROM
Behavioral: non-weight bearing, no range of motion — * 0 weeks to 2 weeks: Posterior plaster slab or cast, non-weightbearing, crutches;
  * At 2 week visit to clinic: Posterior plaster slab or cast removed, staples/stitches removed, BK fibreglass cast or other orthosis applied, with instructions to continue non-weightbearing;
  * At 2 weeks to 6 weeks: Ankle remains immobile and non-weightbearing;
  * After 6 weeks: Begin weightbearing as tolerated. Instructions for limited range of motion to be given, and wean from orthosis.
  Arms: Non-weightbearing no ROM

SUMMARY:
The primary objective of the investigators randomized controlled trial is to determine if early protected weightbearing and ankle range of motion after surgical treatment (open reduction internal fixation - ORIF) for ankle fractures improves the rate of return to work and functional outcome compared to postoperative ankle immobilization in a non-weightbearing cast.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing early weightbearing and mobilization VS immobilization and non-weightbearing after initial treatment of unstable ankle fractures.

The primary objective of our randomized control trial is to determine if early protected weightbearing and ankle range of motion post open reduction internal fixation (ORIF) for unstable ankle fractures improves the rate of return to work and functional outcome compared to postoperative ankle immobilization in a non-weightbearing cast.

Our secondary objective is to determine the rate of adverse events (wound healing, infection, hardware failure) with early weightbearing and ROM comparable to rates with traditional post-op ankle immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral unstable ankle fracture requiring surgical stabilization
* Treatment within two weeks of injury
* Closed or low grade open ankle fracture (grade 1 and/or 2)
* Skeletally mature

Exclusion Criteria:

* Skeletally immature
* Previous ipsilateral ankle surgery
* Bilateral ankle fractures or other major injuries that would affect recovery time
* Grade 3 open fractures
* Inability to co-operate with post-op protocol (advanced dementia, polytrauma patient)
* Non-ambulatory pre injury
* Tibial plafond fractures including articular impaction requiring elevation
* Syndesmosis injury requiring fixation
* Posterior Malleolus fracture - more than 25% of articular surface

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Return to work | 3 months
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work compared to traditional post-op ankle immobilization in a non-weightbearing cast?

SECONDARY OUTCOMES:
Functional outcome and event rate | 2 weeks
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work, functional outcome and rate of adverse events compared to traditional post-op ankle immobilization in a non-weightbearing cast?
Functional outcome and event rate | 6 weeks
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work, functional outcome and rate of adverse events compared to traditional post-op ankle immobilization in a non-weightbearing cast?
Return to work and functional outcome | 9 weeks
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work, functional outcome and rate of adverse events compared to traditional post-op ankle immobilization in a non-weightbearing cast?
Return to work and functional outcome | 6 months
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work, functional outcome and rate of adverse events compared to traditional post-op ankle immobilization in a non-weightbearing cast?
Return to work and functional outcome | 12 months
  Does early weightbearing and ankle range of motion post open reduction internal fixation for unstable ankle fractures improve the rate of return to work, functional outcome and rate of adverse events compared to traditional post-op ankle immobilization in a non-weightbearing cast?

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jenkinson, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre; Hans Kreder, MD,MPH,FRCSC, Study Chair — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hopspital, Toronto, Ontario

REFERENCES:
- [Background] Ahl T, Dalen N, Lundberg A, Bylund C. Early mobilization of operated on ankle fractures. Prospective, controlled study of 40 bimalleolar cases. Acta Orthop Scand. 1993 Feb;64(1):95-9. doi: 10.3109/17453679308994541. PMID 8451961
- [Background] Ahl T, Dalen N, Selvik G. Ankle fractures. A clinical and roentgenographic stereophotogrammetric study. Clin Orthop Relat Res. 1989 Aug;(245):246-55. PMID 2502344
- [Background] Cimino W, Ichtertz D, Slabaugh P. Early mobilization of ankle fractures after open reduction and internal fixation. Clin Orthop Relat Res. 1991 Jun;(267):152-6. PMID 2044269
- [Background] Gul A, Batra S, Mehmood S, Gillham N. Immediate unprotected weight-bearing of operatively treated ankle fractures. Acta Orthop Belg. 2007 Jun;73(3):360-5. PMID 17715727
- [Background] Egol KA, Dolan R, Koval KJ. Functional outcome of surgery for fractures of the ankle. A prospective, randomised comparison of management in a cast or a functional brace. J Bone Joint Surg Br. 2000 Mar;82(2):246-9. PMID 10755435
- [Background] Honigmann P, Goldhahn S, Rosenkranz J, Audige L, Geissmann D, Babst R. Aftertreatment of malleolar fractures following ORIF -- functional compared to protected functional in a vacuum-stabilized orthesis: a randomized controlled trial. Arch Orthop Trauma Surg. 2007 Apr;127(3):195-203. doi: 10.1007/s00402-006-0255-x. Epub 2006 Dec 30. PMID 17195934
- [Background] Lehtonen H, Jarvinen TL, Honkonen S, Nyman M, Vihtonen K, Jarvinen M. Use of a cast compared with a functional ankle brace after operative treatment of an ankle fracture. A prospective, randomized study. J Bone Joint Surg Am. 2003 Feb;85(2):205-11. doi: 10.2106/00004623-200302000-00004. PMID 12571295
- [Background] Lin CW, Moseley AM, Refshauge KM. Rehabilitation for ankle fractures in adults. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005595. doi: 10.1002/14651858.CD005595.pub2. PMID 18646131
- [Background] Nilsson G, Jonsson K, Ekdahl C, Eneroth M. Outcome and quality of life after surgically treated ankle fractures in patients 65 years or older. BMC Musculoskelet Disord. 2007 Dec 20;8:127. doi: 10.1186/1471-2474-8-127. PMID 18096062
- [Background] Obremskey WT, Brown O, Driver R, Dirschl DR. Comparison of SF-36 and Short Musculoskeletal Functional Assessment in recovery from fixation of unstable ankle fractures. Orthopedics. 2007 Feb;30(2):145-51. doi: 10.3928/01477447-20070201-01. PMID 17323637
- [Background] Olerud C, Molander H. A scoring scale for symptom evaluation after ankle fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):190-4. doi: 10.1007/BF00435553. PMID 6437370
- [Background] Petrisor BA, Poolman R, Koval K, Tornetta P 3rd, Bhandari M; Evidence-Based Orthopaedic Trauma Working Group. Management of displaced ankle fractures. J Orthop Trauma. 2006 Jul;20(7):515-8. doi: 10.1097/00005131-200608000-00012. PMID 16891946
- [Background] Shimamura Y, Kaneko K, Kume K, Maeda M, Iwase H. The initial safe range of motion of the ankle joint after three methods of internal fixation of simulated fractures of the medial malleolus. Clin Biomech (Bristol). 2006 Jul;21(6):617-22. doi: 10.1016/j.clinbiomech.2005.12.018. Epub 2006 Feb 24. PMID 16500006
- [Background] Simanski CJ, Maegele MG, Lefering R, Lehnen DM, Kawel N, Riess P, Yucel N, Tiling T, Bouillon B. Functional treatment and early weightbearing after an ankle fracture: a prospective study. J Orthop Trauma. 2006 Feb;20(2):108-14. doi: 10.1097/01.bot.0000197701.96954.8c. PMID 16462563
- [Background] Sondenaa K, Hoigaard U, Smith D, Alho A. Immobilization of operated ankle fractures. Acta Orthop Scand. 1986 Feb;57(1):59-61. doi: 10.3109/17453678608993217. PMID 3083644
- [Background] Strauss EJ, Egol KA. The management of ankle fractures in the elderly. Injury. 2007 Sep;38 Suppl 3:S2-9. doi: 10.1016/j.injury.2007.08.005. PMID 17723786
- [Background] van Laarhoven CJ, Meeuwis JD, van der WerkenC. Postoperative treatment of internally fixed ankle fractures: a prospective randomised study. J Bone Joint Surg Br. 1996 May;78(3):395-9. PMID 8636173
- [Background] Vioreanu M, Dudeney S, Hurson B, Kelly E, O'Rourke K, Quinlan W. Early mobilization in a removable cast compared with immobilization in a cast after operative treatment of ankle fractures: a prospective randomized study. Foot Ankle Int. 2007 Jan;28(1):13-9. doi: 10.3113/FAI.2007.0003. PMID 17257532
- [Background] Siddique Amir, Prasad C.V.R, O'Connor D. Early Active Mobilization Versus Cast Immobilization in Operatively Treated Ankle Fractures. European Journal of Trauma 2005 No4 (31): 398-400
- [Background] Kreder, Hans What is the Role of